CLINICAL TRIAL: NCT02580864
Title: Predictive Factors of Anti-TNFalfa-induced Deep Remission in Crohn's Disease
Brief Title: Bologna IBD Markers
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 13.27.NIHS
Record Dates: First submitted 2015-09-16; First posted 2015-10-20 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, biopsy and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBD patients: 120 adult patients (Caucasian, male/female,18-65 years old) with moderate-severe active Crohns disease (220≤ CDAI ≤450; blood CRP ≥5 mg/L and/or fecal calprotectin ≥250mg/L) and with indication for anti-TNF therapy according to the normal clinical practice
- No-IBD patients: 30 no-IBD controls with no GI disorders, as defined by medical history and standard clinical chemistry values, afferent to the out-patient clinic

SUMMARY:
Individuate possible predictive factors of anti-TNFalfa-induced deep remission in Crohn's disease.

DETAILED DESCRIPTION:
This trial will be exploratory, open in vitro study on human tissues. 120 patients will be enrolled (Caucasian, male/female,18-65 years old) with moderate-severe active Crohns disease and with indication for anti-TNF therapy according to the normal clinical practice.

Simultaneously, 30 no-IBD controls with no GI disorders, as defined by medical history and standard clinical chemistry values, afferent to the out-patient clinic will be enrolled.

ELIGIBILITY:
Main Inclusion Criteria for IBD patients:

* Adult patients (Caucasian)
* Moderate-severe active Crohns disease (220≤ CDAI ≤450; blood CRP ≥5 mg/L and/or fecal calprotectin ≥250mg/L)
* Indication for anti-TNF therapy according to the normal clinical practice
* Informed consent signed

Main Exclusion Criteria for IBD patients:

* Changes of Crohns disease treatment gastrointestinal medication (including corticosteroids) within the previous 2 weeks prior to enrollment
* Pregnant or breast-feeding (at index date) female patients

Main Inclusion Criteria for no-IBD controls:

* No-IBD adult controls (Caucasian) with no GI disorders, as defined by medical history and standard clinical chemistry values, afferent to the out-patient clinic
* Informed consent signed

Main Exclusion criteria for no-IBD controls:

* Medical history of digestive diseases
* Digestive, renal or metabolic disease, as determined by the medical visit and sa blood chemistry analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 adult patients with moderate-severe active Crohns disease with indication for anti-TNF therapy according to the normal clinical practice
  30 no-IBD controls with no GI disorders, as defined by medical history and standard clinical chemistry values, afferent to the out-patient clinic
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of IBD patients in clinical remission at 12 months | 12 months
  * Subjects without intestinal ulceration at endoscopy at 12 months
  * Subjects with CDAI score below 150 from baseline to 12 months
  * Subjects with blood CRP value below 0.8 mg/dL from baseline to 12 months
  * Subjects with stool calprotectin value below 50ug/g from baseline to 12 months
  * Through analysis of metabonomics on biopsies, blood, urine and stools
  * Through analysis of blood genotyping
  * Through analysis of gut microbiota composition

SECONDARY OUTCOMES:
Number of IBD patients requiring an escalation treatment to be in clinical remission at 12 months | Baseline vs Baseline + 12 months
  * Subjects without intestinal ulceration at endoscopy at 12 months
  * Subjects with CDAI score below 150 from baseline to 12 months
  * Subjects with blood CRP value below 0.8 mg/dL from baseline to 12 months
  * Subjects with stool calprotectin value below 50ug/g from baseline to 12 months
  * Through analysis of metabonomics on biopsies, blood, urine and stools
  * Through analysis of blood genotyping
  * Through analysis of gut microbiota composition
Assess phenotypic traits between IBD patients in clinical remission at 12 months and non-IBD subjects | Baseline vs Baseline + 12 months
  * Through analysis of metabonomics on blood, urine and stools
  * Through analysis of gut microbiota composition
  * Through clinical nutritional status in IBD patients compared to non-IBD subjects
Assess healthy intra-individual variability of gut microbial activity and dietary behavior in relation to disease development and management | Baseline
  * Through analysis of gut microbiota composition
  * Through clinical nutritional status

CONTACTS AND LOCATIONS:
Locations (1):
- Bologna University, Bologna, Italy

REFERENCES:
- [Derived] Rizzello F, Gionchetti P, Spisni E, Saracino IM, Bellocchio I, Spigarelli R, Collini N, Imbesi V, Dervieux T, Alvisi P, Valerii MC. Dietary Habits and Nutrient Deficiencies in a Cohort of European Crohn's Disease Adult Patients. Int J Mol Sci. 2023 Jan 12;24(2):1494. doi: 10.3390/ijms24021494. PMID 36675009